CLINICAL TRIAL: NCT03690180
Title: Hypomagnesemia as a Marker of Diabeteiv Nephropathy
Brief Title: Hypomagnesemia and Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of Medicine,Faculty of Medicine,Fayoum university, Fayoum University
Other Study IDs: VCG5
Record Dates: First submitted 2018-03-31; First posted 2018-10-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics with microalbuminuria: Diabetics with micro albuminuria will be subjected to full clinical examination.
  Measurement of weight, height, waist, hip and calculation of BMI and waist hip ratio,laboratory assessment of serum creatinine,HbA1C,magnesium and urinary albumin creatinine ratio
  Interventions: Diagnostic Test: serum magnesium
- Diabetics with normal albuminuria: Diabetics with micro albuminuria will be subjected to full clinical examination.
  Measurement of weight, height, waist, hip and calculation of BMI and waist hip ratio,laboratory assessment of serum creatinine,HbA1C,magnesium and urinary albumin creatinine ratio
  Interventions: Diagnostic Test: serum magnesium

INTERVENTIONS:
Diagnostic Test: serum magnesium — assessment of serum magnesium in all patients

SUMMARY:
To find if there is a corrolatation between Microalbuminurea and diabetic retinopathy, in daibetic patients

DETAILED DESCRIPTION:
40 Daibetic patients with microalbuminurea will be subjeted to full clinical examination and fundus examination,20 control diabetics with out microalbuminurea will also be included for comparison,patients will be selected from the outpatient clinic 0f fayoum university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics on oral treatment,diabetics on insulin

Exclusion Criteria:

* Healthy volunteers,,hypertensive patients with normal blood glucose

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients following up in out patient clinic of diabetes and endocrine ,Fayoum university Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Decrease in serum magnesium | One month
  statistical significant change in serum magnesium in diabetics with microalbuminuria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Fayoum univesity, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided